CLINICAL TRIAL: NCT03100916
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 690517 in Healthy Male Subjects (Single-blind, Partially Randomised, Placebo-controlled Within Dose Groups) and Effect of Food on the Bioavailability of BI 690517 (Openlabel, Randomised, Two-way Cross-over)
Brief Title: This Study Tests How Different Doses of BI 690517 Are Taken up in the Body of Healthy Men. The Study Also Looks at How Food Influences the Amount of BI 690517 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1378-0002; 2017-000104-18 (EudraCT Number)
Record Dates: First submitted 2017-03-31; First posted 2017-04-04 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Ranging Arm (Experimental)
  Interventions: Drug: BI 690517; Drug: Placebo
- Food Effect arm (Experimental)
  Interventions: Drug: BI 690517 (Reference); Drug: BI 690517

INTERVENTIONS:
Drug: BI 690517 — once daily
  Other Names: Vicadrostat
  Arms: Dose Ranging Arm
Drug: Placebo — once daily
  Arms: Dose Ranging Arm
Drug: BI 690517 (Reference) — Fasting
  Other Names: Vicadrostat
  Arms: Food Effect arm
Drug: BI 690517 — Non- fasting
  Other Names: Vicadrostat
  Arms: Food Effect arm

SUMMARY:
The primary objective of the trial is to investigate the safety and tolerability of BI 690517 in healthy male subjects following oral administration of multiple rising doses over 14 days (MRD part).

Secondary objectives for the MRD part are the exploration of PK (Pharmacokinetic(s)), including dose proportionality, as well as investigation of linearity and PD (Pharmacodynamic(s)) of BI 690517 after multiple dosing.

For the FE (food effect) part, the secondary objective is to investigate the relative bioavailability of BI 690517 under fasted conditions (Reference, R) compared to BI 690517 (single dose) after a high fat high caloric breakfast (Test, T).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP(Blood Pressure), PR (Pulse Rate)), 12-lead ECG (Electrocardiogram), and clinical laboratory tests
* Age of 18 to 50 years (incl.)
* BMI(Body Mass Index) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and local legislation
* Willingness to comply with contraception requirements. Subjects who are sexually active must use adequate contraception with their female partner throughout the study and until one month after the last administration of trial medication. Adequate methods are:

  * Sexual abstinence or
  * A vasectomy performed at least 1 year prior to screening in combination with a barrier method (condom) or
  * Surgical sterilisation (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner or
  * The use of condoms, if the female partner uses an adequate contraception method in addition, e.g., intrauterine device (IUD), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration, or barrier method (e.g. diaphragm with spermicide) Unprotected sexual intercourse with a female partner is not allowed throughout the study and until one month after the last administration of trial medication.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts; orthostatic dysregulation identified during screening or on Day 1)
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients or Synacthen®), previous diagnostic test with Synacthen®
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Values for serum sodium and potassium outside normal range at screening
* Male subjects with WOCBP partner who are unwilling to use male contraception (condom or sexual abstinence) from the first administration of trial medication until 30 days after last administration of trial medication

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
[N (%)] of subjects with drug-related Adverse Events | Day 30
  [N (%)] of subjects with drug-related Adverse Events

SECONDARY OUTCOMES:
AUCtau,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval tau after administration of the first dose [AUCtau,1 will be AUC0-24]) | 0-24 hours
  AUCtau,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval tau after administration of the first dose [AUCtau,1 will be AUC0-24])
Cmax (maximum measured concentration of the analyte in plasma) (After the first dose)(Multiple rising dose part) | up to 24 hours
  Cmax (maximum measured concentration of the analyte in plasma) (After the first dose)(Multiple rising dose part)
AUCtau,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval tau)(After the last dose)(Multiple rising dose part) | 312 - 360 hours
  AUCtau,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval tau)(After the last dose)(Multiple rising dose part)
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval tau)(After the last dose)(Multiple rising dose part) | after 312 hours and up to 360 hours
  Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval tau)(After the last dose)(Multiple rising dose part)
Cmax (maximum measured concentration of the analyte in plasma) (Food effect part) | Up to 48 hours
  Cmax (maximum measured concentration of the analyte in plasma) (Food effect part)
AUC0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 48 hours
  AUC0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
AUC0- tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | Up to 48 hours
  AUC0- tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany